CLINICAL TRIAL: NCT03871218
Title: Evaluation of the Effect of Hyaluronic Acid Application on the Healing of the Donor and Recipient Sites After Free Gingival Graft With Laser Doppler Flowmetry
Brief Title: Effect of Hyaluronic-acid on the Healing After Free Gingival Graft
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Zeynep Turgut Çankaya, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19.04.2017 08/14
Record Dates: First submitted 2019-03-10; First posted 2019-03-12 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2017-04

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: After FGG was taken from the donor region in the TG, sterile gauze was applied with moderate pressure for 2 minutes, and HA was applied topically after the bleeding stopped. In the TG, HA was applied to the entire recipient bed before suturing the graft taken from the palatial mucosa to the recipient site. In the control group (CG), HA was not applied to the recipient or the donor site.
Who Masked: Outcomes Assessor
Masking Description: examiner blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Active Comparator): Hyaluronic acid application group. After FGG was taken from the donor region in the TG, sterile gauze was applied with moderate pressure for 2 minutes, and HA was applied topically after the bleeding stopped. The cross-linked HA package containing 20 mg/ml Na-hyaluronate, stored at room temperature, was opened, and the protective cap of the syringe was removed.
  Interventions: Biological: Hyaluronic acid group
- Control Group (No Intervention): In the control group (CG), HA was not applied to the recipient or the donor site.

INTERVENTIONS:
Biological: Hyaluronic acid group — Applicaton of topical Hyaluronic acid
  Arms: Test Group

SUMMARY:
This study evaluated the effect of topical hyaluronic acid (HA) application on free gingival graft (FGG) donor and recipient sites during the early wound healing period with laser Doppler flowmetry (LDF) and to investigate the effect of HA application on the dimensional change of the graft.Participants were randomly classified into the test group (TG) and control group (CG). HA was applied to both donor and recipient sites in 20 patients who formed the TG, whereas HA was not applied to the 20 patients who formed the CG.

DETAILED DESCRIPTION:
The healing of a transplanted tissue depends on the formation of blood support between the donor and recipient sites.

Hyaluronic acid (HA) is a biomaterial that creates a favorable environment for wound healing due to its unique hydroscopic and viscoelastic properties, and it is important for wound healing activities.HA induces angiogenesis following degradation and improves the wound healing environment.HA supports a mechanism that induces proliferation of capillaries, and components produced after HA degradation increase vascularization.Laser Doppler flowmetry (LDF) technique is frequently used in the field of plastic surgery for monitoring microvascular blood flow to detect insufficient circulation in the skin transplants and flaps in the early period and to thereby prevent and predict possible surgical complications.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed inadequate attached gingiva

Exclusion Criteria:

* Smoking

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
blood perfusion value in the recipient bed | on day 4
  The comparison of blood perfusion value in the recipient bed between the TG and CG on day 4

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Turgut Çankaya, Principal Investigator — Gazi University
Locations (1):
- Gazi University Faculty of Dentistry Department of Periodontology, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No